CLINICAL TRIAL: NCT02159430
Title: Hereditary AngioEdema, Neurobiology and Psychopathology
Acronym: HAENP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Catania (Other)
Responsible Party: Principal Investigator, Prof. Eugenio Aguglia, Full Professor of Psychiatry, University Hospital, Catania
Other Study IDs: UHCatania1
Record Dates: First submitted 2014-06-05; First posted 2014-06-10 (Estimated); Last update posted 2014-06-10 (Estimated); Status verified 2014-06

CONDITIONS: Hereditary AngioEdema; Anxiety; Depression
MeSH Terms: conditions — Angioedemas, Hereditary; Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HereditaryAngioEdema: Patients from the Eastern Sicily HAE register
  Interventions: Other: Clinical and psychopathological assessment of HAE patients

INTERVENTIONS:
Other: Clinical and psychopathological assessment of HAE patients

SUMMARY:
Since 1963 Hereditary AngioEdema (HAE) is considered an autosomal dominant disorder (Donaldson and Evans), characterized by a quantitative and/or qualitative deficit of C1 esterase inhibitor (C1-INH), which affects approximately 1:50.000 individuals in the general population. From this period the link between HAE and psychiatry was interrupted, however genetic issues could not comprehensively explain the clinical evolution of the disease. Clinical studies show an evident gap between genotype and phenotype of HAE. For this still controversial question, we have designed this cross-sectional study in order to establish the relationship between HAE clinical manifestations and neurobiological/psychopatological parameters.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of HAE

Exclusion Criteria:

* Current pharmacological treatment including ACE-inhibitors, ACE inhibitors, glucocorticoids, oestroprogestative, psychotropic drugs, drugs acting on the immune system (15 days before), anesthetics (in the previous three months).
* Inflammation / infection (eg, chronic inflammatory diseases, acute) in the last 15 days.
* Ongoing allergies.
* Night work over the past 15 days.
* Vigorous physical activity or alcohol consumption (the day before the assessment).
* Women in follicular phase of menstrual cycle.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This population-based cross-sectional study will include all Hereditary AngioEdema (HAE) patients from the Eastern Sicily HAE register.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-02 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Multivariate linear regression analysis of HAE clinical status and psychometric parameters | First assessment

CONTACTS AND LOCATIONS:
Locations (1):
- UOPI of psychiatry - Department of clinical and molecular biomedicine - AOU Policlinico-Vittorio Emanuele, Catania, Catania, Italy